CLINICAL TRIAL: NCT05405946
Title: Computerized Cognitive Remediation Therapy in Adolescents With a First Psychotic Episode: Randomized Controlled Trial
Brief Title: Computerized Cognitive Remediation Therapy in Adolescents With a First Psychotic Episode
Acronym: CCRT2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSJD-CCRT-2019; PIC-99-19 (Other: CEIM Certificate)
Record Dates: First submitted 2022-01-24; First posted 2022-06-06 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Early-onset Schizophrenia; Psychotic Disorders; Cognitive Remediation Therapy; Cognition
Keywords: Early-onset; Psychotic Disorders; Cognitive Remediation Therapy; CRT; Cognition; Functional Outcome; Adolescent
MeSH Terms: conditions — Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The group will be randomized as parallel groups. CCRT Group in comparison with TAU Group. Randomization will be performed using permuted blocks with a fixed size of 8 patients assigned in a relationship 4:4 according to the computerized assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Cognitive Remediation Intervention and Treatment as Usual (CCRT+TAU) (Experimental): Participants with a diagnosis of schizophrenia / schizoaffective disorder undergo Computerized CRT and the usual treatment.
  Three evaluations are carried out, each one divided into two sessions: an evaluation before the start of treatment, a second evaluation after finishing the Computerized CRT (after 40 sessions), and a third evaluation (follow-up) 6 months after finishing the Computerized CRT.
  Interventions: Behavioral: Computerized Cognitive Remediation Therapy; Other: Treatment as Usual
- Treatment as Usual (TAU) (Active Comparator): Participants with a diagnosis of schizophrenia / schizoaffective disorder undergo the usual treatment.
  Two evaluations will be carried out, also divided into two sessions: a first baseline evaluation and a second evaluation 5 months later, after receiving the usual treatment. After this second evaluation, the Computerized CRT is then started to guarantee ethics in all patients.
  The evaluation is not carried out at 6 months since they will also have received the intervention.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Computerized Cognitive Remediation Therapy — Sessions of 45 minutes will be developed 2 times a week, for 4-5 months (performing a total of 40 sessions). The sessions will be led by an experienced clinician with psychotic patients, and trained for the management of CCRT. Each intervention session will be individualized according to the results of the evaluation tests and the computerized program itself will adapt the difficulty of the tasks according to the performance of each patient.
  The cognitive remediation NeuroPersonalTrainer platform includes two rehabilitation modules: the cognition module that includes attention, memory and executive functions with different levels of complexity and the Social Cognition module which allows working on different aspects of emotional processing, theory of mind and cognitive biases through 43 tasks based on multiple multimedia materials.
  Other Names: CCRT
  Arms: Computerized Cognitive Remediation Intervention and Treatment as Usual (CCRT+TAU)
Other: Treatment as Usual — Patients receiving TAU include psychoeducation about the disorder, psychiatric visits, and follow-up and review of drug treatment. In addition, they make individual visits with psychology, nursing and / or social work. In all cases, patients are treated in outpatient clinics.
  Other Names: TAU

SUMMARY:
Cognitive deficits (CD) are considered one of the essential characteristics in psychotic disorders and occur throughout the course of the disease, being a key characteristic in the evolution of the disease and in the functionality and prognosis of patients. Intervening in the early stages of the disease and specifically in adolescence, a period of high brain plasticity can reduce disabilities in adulthood associated with early-onset psychosis. The objective of this study is to assess the efficacy of cognitive rehabilitation therapy in adolescents with a first psychotic episode, comparing two groups of these patients: a first group (CCRT) will carry out 40 sessions of a computerized cognitive remediation therapy with the usual treatment too, and a second group will perform only the usual treatment (TAU). The main hypothesis is that the CCRT group will present a significant improvement in verbal memory, visual attention, executive function, and social cognition and will present better global functioning compared to the TAU group.

DETAILED DESCRIPTION:
Cognitive deficits (DC) are considered one of the essential features in psychotic disorders and occur throughout the course of the disease. Recent meta-analyses have shown that cognitive remediation therapy can reduce DCs in basic cognitive processes such as attention, memory, and problem solving and can have an impact on social functioning.

The aim of this study is to evaluate the effectiveness of a computerized cognitive remediation intervention in cognitive and functional improvement in patients with a first psychotic episode that is psychopathologically stable but presents cognitive impairment.

The hypotheses that are raised are:

1. In relation to the cognitive field. Participants in the computerized cognitive remediation therapy + treatment as usual (CCRT) group versus the participants in the treatment as usual (TAU) group are expected to improve in (evaluated by MATRICS):

   1. Verbal memory
   2. Visual attention
   3. Executive function
   4. Social cognition
2. In relation to other symptoms. Participants in the CCRT group versus the participants in the TAU group are expected to:

   1. Present better Global Functioning evaluated through C-GAS.

      Parallel groups will be compared with patients between 12 and 18 years of age diagnosed with schizophrenia / schizoaffective recruited at the Hospital Sant Joan de Déu Barcelona. A total of 50 randomly distributed patients will be included (n = 25 CCRT; n = 25 TAU). CCRT group will perform a total of 40 computerized cognitive remediation (cCR) sessions through the NeuroPersonalTrainer program in addition to the treatment as usual, and TAU group will perform only the treatment as usual. An evaluation will be performed before the start of treatment, a second evaluation after the end of the 40cCRsessions/ TAU, and a third evaluation (follow-up) 6 months after the end of the 40cCRsessions.

      Data Management

      The aforementioned variables will be collected on the one hand in paper format, in a data collection notebook created by ADHOC for the study that will be kept with a key and the data in electronic format, derived from the computerized programs and tests will be stored with a password, all of this under the responsibility of the principal investigator. The monitoring plan consists in that each visit made to carry out the study will be recorded in the participant's clinical history and the variables of clinical or neuropsychological interest will be included in the history and in a way that can be accessed to verify the data. Verification of all the data of each participant will be carried out once the study has been completed by the participant and the data collection has been completed and all the participant's data has been coded. Data that cannot be recovered will be coded as "missing" and participants who could not be tracked as "drop-outs".

      The data of each participant will be coded and included in a database for later analysis. Data that could lead to the identification of the participant will not be stored in the database. No information of any kind to identify the participants will be included. Only the study doctor and his collaborators will be able to relate the data collected in the study with his medical history.

      No adverse effects are expected as it is a protocol that does not include drugs or invasive procedures. In the case of detecting an adverse effect, it would be notified and coded in the database.

      Statistical analysis

      The group will be randomized as follows: parallel, CCRT Group compared to TAU Group. Randomization will be performed using permuted blocks with a fixed size of 8 patients assigned a 4: 4 ratio according to computerized allocation i is done blindly. Randomization is performed by an outside person to whom the program applies. Following the CONSORT statement for controlled trials (Moher et al. 2010), the intention-to-treat analysis will be used. This consists of the comparison of the CCRT Group, including all patients, as originally assigned after randomization. The analysis of the missing and drop-outs will also be carried out according to the CONSORT statement. An analysis of the descriptive and contingency tables will be carried out. Tests will be carried out to evaluate the normality of the results through the Kolmogorov-Smirnov test. For variables with a normal distribution, Student's t-test will be applied and non-parametric tests (U-Mann Witney) will be applied for results without normal distribution.

      For the evaluation of the pre-post differences, repeated measures analysis of variance (ANOVA) designed with the CCRT Group versus TAU Group condition will be used as the independent variable and the baseline and post-treatment evaluations as the time points. An analysis of covariance with repeated measures (ANCOVA) will be performed, including potentials as covariates. The effect size for calculating changes in scores will be calculated in 2 complementary groups in two ways. Eta partial squared (h2p) will be used to calculate the effect size of the scores between baseline and post-treatment evaluations. The effect size of the number needed to treat (NNT) will also be calculated since it is a clinically significant measure that indicates the number of people who would need to be treated to achieve a specific therapeutic goal. Furthermore, it will be determined if the cognitive changes are reliable using TAU Group test-re-test reliability coefficients in order to calculate the standard error of measurement according to Medalia (2005). CCRT Group patients whose score changes to a coefficient value of 1.64 or higher (90% CI) will be identified as a reliable improvement. Finally, the use of repeated measures ANOVA will be used to assess changes from baseline to 3-month follow-up in CCRT Group, with baseline and follow-up as time points. Logistic regression models will also be included to study dichotomous variables in the event that the bivariate analysis has been significant. For the statistical analysis, the statistical package STATA 12 will be used.

      Data codebook

      Code=RHC_0XX Age=Date of birth Sex=Sex

      N_Sessions=Sessions performed

      Peduc=paternal education level Meduc=maternal education level Poccup=paternal occupation Moccup=maternal occupation residence=place of residence kindh=kind of house Npobl=nº hab poblacion Npersh=number of persons at home SES=socioeconomic status F_Psq_history=Family Psyquiatric History

      OSC=Obstetric Risk perinatal=perinatal history psychomot=psychomotor development language=language development read_write=reading and writing development Psq_history= Personal Psychiatric History Psq_age=age first contact mental health service Psq_pharma=history of pharmacological treatment Psq_psychology=history of psychological treatments Psq_1HOSP_age=age of first hospitalization Psq_1HOSP_days=days first hospitalization Medical_history=relevant medical history academic_rep=repetition of academic year course=academic level freq_subs_lifec= maximum frequency of café throughout life freq_subs_3m= frequency of café last 3 months

      K-SADS-PL-5: Psychopathology PANS-PS_0: Positive symptoms basal PANS-PS_40s: Positive symptoms 40 sessions follow-up PANS-PS_6m: Positive symptoms 6 months follow-up PANS-NS_0: Negative symptoms basal PANS-NS_40s: Negative symptoms 40 sessions follow-up PANS-DS_6m: Negative symptoms 6 months follow-up PANS-DS_0: Disorganization symptoms basal PANS-DS_40s: Disorganization symptoms 40 sessions follow-up PANS-DS_6m: Disorganization symptoms 6 months follow-up GAF_0= Global Functioning basal GAF_40s= Global Functioning 40 sessions follow-up GAF_6m= Global Functioning 6 months follow-up

      W_V_Pd=Vocabulary direct W_V_T= Vocabulary t-score W_C_Pd= Block Design direct W_C_T= Block Design t-score W_S_Pd= Similarities direct W_S_T= Similarities t-score W_M_Pd=Matrix reasoning direct W_M_T Matrix reasoning t-score W_B_Pd=Figure Weights direct W_B_T=Figure Weights t-score ICV_Pe= Verbal Comprehension ICV_CI= Verbal Comprehension Index IFR_Pe= Fluid Reasoning IFR_CI= Fluid Reasoning Index ICG_Pe= General Ability ICG_CI= General Ability Index W_DT_Pd_0= working memory Digit span direct W_DT_T_0= working memory Digit span t-score W_Dd_Pd_0= working memory direct Digit span direct W_Dd_Pd_0= working memory direct Digit span t-score W_Di_Pd_0= working memory indirect Digit span direct W_Di_Pd_0= working memory indirect Digit span t-score W_CN_Pd_0= Processing Speed coding direct W_CN_Pd_0= Processing Speed coding t-score W_LN_Pd_0= working memory Letter-number sequencing direct W_LN_T_0= working memory Letter-number sequencing t-score W_DT_Pd_40s= working memory Digit span direct 40 sessions follow-up W_DT_T_40s = working memory Digit span t-score 40 sessions follow-up W_Dd_Pd_40s = working memory direct Digit span direct 40 sessions follow-up W_Dd_Pd_40s = working memory direct Digit span t-score 40 sessions follow-up W_Di_Pd_40s = working memory indirect Digit span direct 40 sessions follow-up W_Di_Pd_40s = working memory indirect Digit span t-score 40 sessions follow-up W_CN_Pd_40s = Processing Speed coding direct 40 sessions follow-up W_CN_Pd_40s = Processing Speed coding t-score 40 sessions follow-up W_LN_Pd_40s = working memory Letter-number sequencing direct 40 sessions follow-up W_LN_T_40s = working memory Letter-number sequencing t-score 40 sessions follow-up W_DT_Pd_6m= working memory Digit span direct 6 months follow-up W_DT_T_6m= working memory Digit span t-score 6 months follow-up W_Dd_Pd_6m= working memory direct Digit span direct 6 months follow-up W_Dd_Pd_6m= working memory direct Digit span t-score 6 months follow-up W_Di_Pd_6m= working memory indirect Digit span direct 6 months follow-up W_Di_Pd_6m= working memory indirect Digit span t-score 6 months follow-up W_CN_Pd_6m= Processing Speed coding direct 6 months follow-up W_CN_Pd_6m= Processing Speed coding span t-score 6 months follow-up W_LN_Pd_6m= working memory Letter-number sequencing direct 6 months follow-up W_LN_T_6m= working memory Letter-number sequencing t-score 6 months follow-up CPT_CI_0=Attention basal CPT_CI_40s=Attention 40 sessions follow-up CPT_CI_RP=Attention 6 months follow-up CPT_O_0= Attention, omissions basal CPT_O_40s =Attention, omissions 40 sessions follow-up CPT_O_RP=Attention, omissions 6 months follow-up CPT_C_0= Attention, commissions basal CPT_C_40s =Attention, commissions 40 sessions follow-up CPT_C_RP=Attention, commissions 6 months follow-up CPT_HRT_0= Attention, reaction time basal CPT_HRT_40s =Attention, reaction time 40 sessions follow-up CPT_HRT_RP=Attention, reaction time 6 months follow-up CPT_D_0= Attention, detectability basal CPT_D_40s =Attention, detectability 40 sessions follow-up CPT_D_RP=Attention, detectability 6 months follow-up CPT_V_0= Attention, variability basal CPT_V_40s =Attention, variability 40 sessions follow-up CPT_V_RP=Attention, variability 6 months follow-up TMT-A_Pd_0=Processing Speed TMT-A, direct score basal TMT-A_Pd_40s=Processing Speed TMT-A, direct score 40 sessions follow-up TMT-A_Pd_RP=Processing Speed TMT-A, direct score , 6 months follow-up TMT-A_T_0=Processing Speed TMT-A, t-score basal TMT-A_T_40s=Processing Speed TMT-A, t-score, 40 sessions follow-up TMT-A_T_6m=Processing Speed TMT-A, t-score, 6 months follow-up TMT-B_Pd_0=executive functions TMT-B, direct score basal TMT-B_Pd_40s=executive functions TMT-B, direct score 40 sessions follow-up TMT-B_Pd_RP=executive functions TMT-B, direct score , 6 months follow-up TMT-B_T_0=executive functions TMT-B, t-score basal TMT-B_T_40s=executive functions TMT-B, t-score, 40 sessions follow-up TMT-B_T_6m=executive functions TMT-B, t-score, 6 months follow-up HVLT_Pd_0=Long term Verbal Memory, direct, basal HVLT_Pd_40s =Long term Verbal Memory, direct, 40 sessions follow-up HVLT_Pd_6m =Long term Verbal Memory, direct, 6 months follow-up HVLT_T_0=Long term Verbal Memory, t-score basal HVLT_T_40s =Long term Verbal Memory t-score 40 sessions follow-up HVLT_T_6m =Long term Verbal Memory t-score 6 months follow-up HVLT_Pd_0=Verbal Memory Learning, direct, basal HVLT_Pd_40s =Verbal Memory Learning, direct, 40 sessions follow-up HVLT_Pd_6m =Verbal Memory Learning, direct, 6 months follow-up HVLT_T_0=Verbal Memory Learning, t-score basal HVLT_T_40s =Verbal Memory Learning, t-score 40 sessions follow-up HVLT_T_6m =Verbal Memory Learning, t-score 6 months follow-up Rey_CQ_0= Copy Quality Visual Memory basal Rey_CQ_40s = Copy Quality Visual Memory 40 sessions follow-up Rey_CQ_6m = Copy Quality Visual Memory 6 months follow-up Rey _CA_0= Copy Accuracy Visual Memory basal Rey_CA_40s = Copy Accuracy Visual Memory 40 sessions follow-up Rey_CA_6m = Copy Accuracy Visual Memory 6 months follow-up Rey _MQ_0= Memory Quality Visual Memory basal Rey_MQ_40s =Memory Quality Visual Memory 40 sessions follow-up Rey_MQ_6m =Memory Quality Visual Memory 6 months follow-up Rey_MA_0= Memory Accuracy Visual Memory basal Rey_MA_40s =Memory Accuracy Visual Memory 40 sessions follow-up Rey_MA_6m =Memory Accuracy Visual Memory 6 months follow-up WSCT_E_0= executive functions, WSCT total errors basal WSCT_E_40s = executive functions, WSCT total errors 40 sessions follow-up WSCT_E_6m = executive functions, WSCT total errors 6 months follow-up WSCT_PE_0= executive functions, WSCT percentage errors basal WSCT_PE_40s = executive functions, WSCT percentage errors totals 40 sessions follow-up WSCT_PE_6m = executive functions, WSCT percentage errors totals 6 months follow-up WSCT_persev_0= executive functions, WSCT persevering responses basal WSCT_persev_40s = executive functions, WSCT persevering responses 40 sessions follow-up WSCT_persev_6m = executive functions, WSCT persevering responses 6 months follow-up WSCT_Epersev_0= executive functions, WSCT persevering errors basal WSCT_Epersev_40s = executive functions, WSCT persevering errors 40 sessions follow-up WSCT_Epersev_6m = executive functions, WSCT persevering errors 6 months follow-up WSCT_PEpersev_0= executive functions, WSCT percentage persevering errors basal WSCT_PEpersev_40s = executive functions, WSCT percentage persevering errors 40 sessions follow-up WSCT_PEpersev_6m = executive functions, WSCT percentage persevering errors 6 months follow-up WSCT_ENopersev_0= executive functions, WSCT non-persevering errors basal WSCT_ENopersev_40s = executive functions, WSCT non-persevering errors 40 sessions follow-up WSCT_ENopersev_6m = executive functions, WSCT non-persevering errors 6 months follow-up WSCT_PENopersev_0= executive functions, WSCT percentage non-persevering errors basal WSCT_PENopersev_40s = executive functions, WSCT percentage non-persevering errors 40 sessions follow-up WSCT_PENopersev_6m= executive functions, WSCT percentage non-persevering errors 6 months follow-up WSCT_categories_0= executive functions, WSCT categories basal WSCT_categories_40s = executive functions, WSCT categories non-persevering errors 40 sessions follow-up WSCT_categories_6m= executive functions, WSCT categories 6 months follow-up FAS_Pd_0=Processing Speed FAS Word Fluency, direct scores basal FAS_Pd_40s=Processing Speed FAS Word Fluency, direct scores 40 sessions follow-up

      FAS_T_6m=Processing Speed FAS Word Fluency, direct scores 6 months follow-up FAS_T_0=Processing Speed FAS Word Fluency, t-scores basal FAS_T_40s=Processing Speed FAS Word Fluency, t-scores40 sessions follow-up FAS_T_6m=Processing Speed FAS Word Fluency, t-scores 6 months follow-up Semantic_Pd_0=Processing Speed Semantic Word Fluency, direct scores basal Semantic_Pd_40s=Processing Speed Semantic Word Fluency, direct scores 40 sessions follow-up Semantic _Pd_6m=Processing Speed Semantic Word Fluency, direct scores 6 months follow-up Semantic _T_0=Processing Speed Semantic Word Fluency, t-scores basal Semantic _T_40s=Processing Speed Semantic Word Fluency, t-scores 40 sessions follow-up Semantic _T_6m=Processing Speed Semantic Word Fluency, t-scores 6 months follow-up FACES_Pd_0= Social Cognition basal FACES_Pd_40s= Social Cognition 40 sessions follow-up FACES_Pd_6m= Social Cognition 6 months follow-up

ELIGIBILITY:
Inclusion Criteria:

* 1) Age between 12-18 years
* 2) DSM-5 diagnostic criteria for schizophrenia or schizoaffective disorder (F20 or F25, DSM-5) beginning at age 17 or earlier;
* 3) Clinically and pharmacologically stabilized;
* 3) No changes in drug treatment for 6 weeks from baseline assessment;
* 4) Presence of cognitive impairment according to criteria adapted in Penades et al. and following the same criteria in previous studies with similar populations. In this sense, at least one of the following criteria must be present:

  1. 2 discrepant scores (a score is discrepant when the T scores are 1 DE below the patient's estimated IQ
  2. Either a score T below 37 in persevering Wisconsin Card Sorting Test (WCST) errors by Heaton et al. (1981).
* 5) Diagnosis and diagnostic stability verified by a psychiatrist or senior psychologist or member of the research team using the DSM-5 criteria and based on clinical interviews with the patient and his family.

Exclusion Criteria:

* 1) Intellectual disability CI estimated equivalent to or <70);
* 2) Active substance abuse;
* 3) Neurological impairment;
* 4) Have received electro-convulsive therapy in the 6 months prior to treatment;
* 5) Do not sign informed consent.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Global Functioning | 1 week
  T-score, GAF: Global Assesment Functioning-Scale (Endicott et al, 1976) Range: 0 (lowest) to 100 (highest)
Global Functioning | 5 months
  T-score, GAF: Global Assesment Functioning-Scale (Endicott et al, 1976) Range: 0 (lowest) to 100 (highest)
Global Functioning | 11 months
  T-score, GAF: Global Assesment Functioning-Scale (Endicott et al, 1976) Range: 0 (lowest) to 100 (highest)
Long term Verbal Memory | 1 week
  T-score, long term, Hopkins Verbal Learning Test- Revised (HVLT-R; Brandt 1991)
Long term Verbal Memory | 5 months
  T-score, long term, Hopkins Verbal Learning Test- Revised (HVLT-R; Brandt 1991)
Long term Verbal Memory | 11 months
  T-score, long term, Hopkins Verbal Learning Test- Revised (HVLT-R; Brandt 1991)
Verbal Memory, Learning | 1 week
  T-score, learning, Hopkins Verbal Learning Test- Revised (HVLT-R; Brandt 1991)
Verbal Memory, Learning | 5 months
  T-score, learning, Hopkins Verbal Learning Test- Revised (HVLT-R; Brandt 1991)
Verbal Memory, Learning | 11 months
  T-score, learning, Hopkins Verbal Learning Test- Revised (HVLT-R; Brandt 1991)
Attention | 1 week
  Confidence Index, Continuous Performance Test - II (CPT-II; Rosvold, 1956)
Attention | 5 months
  Confidence Index, Continuous Performance Test - II (CPT-II; Rosvold, 1956)
Attention | 11 months
  Confidence Index, Continuous Performance Test - II (CPT-II; Rosvold, 1956)
Long Term Visual Memory | 1 week
  T-score, long term, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991)
Long term Visual Memory | 5 months
  T-score, long term, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991)
Long term Visual Memory | 11 months
  T-score, long term, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991)
Organization Visual Memory | 1 week
  Percentile, organization, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991)
Organization Visual Memory | 5 months
  Percentile, organization, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991)
Organization Visual Memory | 11 months
  Percentile, organization, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991)
Working memory Spatial Span (WISC-V) | 1 week
  T-score, Spatial Span Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014)
Working memory Spatial Span | 1 week
  T-score, Spatial Span Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012)
Working memory Spatial Span (WISC-V) | 5 months
  T-score, Spatial Span Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014)
Working memory Spatial Span | 5 months
  T-score, Spatial Span Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012)
Working memory Spatial Span (WISC-V) | 11 months
  T-score, Spatial Span Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014)
Working memory Spatial Span | 11 months
  T-score, Spatial Span Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012)
Working memory Letter-Number Span (WISC-V) | 1 week
  T-score: Letter-Number Span Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014)
Working memory Letter-Number Span | 1 week
  T-score: Letter-Number Span Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012)
Working memory Letter-Number Span (WISC-V) | 5 months
  T-score: Letter-Number Span Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014)
Working memory Letter-Number Span | 5 months
  T-score: Letter-Number Span Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012)
Working memory Letter-Number Span (WISC-V) | 11 months
  T-score: Letter-Number Span Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014)
Working memory Letter-Number Span | 11 months
  T-score: Letter-Number Span Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012)
Working memory digits (WISC-V) | 1 week
  T-score, Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014)
Working memory digits | 1 week
  T-score, Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
Working memory digits (WISC-V) | 5 months
  T-score, Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
Working memory digits | 5 months
  T-score, Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
Working memory digits (WISC-V) | 11 months
  T-score, Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
Working memory digits | 11 months
  T-score, Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
Social Cognition | 1 week
  Faces Test de Baron-Cohen (Wheelwright y Jolliffe,1997) Range: 0 (lowest) to 28 (highest)
Social Cognition | up to 5 months
  Faces Test de Baron-Cohen (Wheelwright y Jolliffe,1997) Range: 0 (lowest) to 28 (highest)
Social Cognition | 11 months
  Faces Test de Baron-Cohen (Wheelwright y Jolliffe,1997) Range: 0 (lowest) to 28 (highest)
Executive functions, categories | 1 week
  T-score, Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
Executive functions, categories | 5 months
  T-score, Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
Executive functions, categories | 11 months
  T-score, Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
Executive functions, TMT-B | 1 week
  T-score, Trail Making Test: Part B (TMT; Reitan, 1971) Range: 0 (lowest) to 100 (highest)
Executive functions, TMT-B | 5 months
  T-score, Trail Making Test: Part B (TMT; Reitan, 1971) Range: 0 (lowest) to 100 (highest)
Executive functions, TMT-B | 11 months
  T-score, Trail Making Test: Part B (TMT; Reitan, 1971) Range: 0 (lowest) to 100 (highest)
Processing Speed TMT-A | 1 week
  T-score, Trail Making Test: Part A (TMT; Reitan, 1971) Range: 0 (lowest) to 100 (highest)
Processing Speed TMT-A | 5 months
  T-score, Trail Making Test: Part A (TMT; Reitan, 1971) Range: 0 (lowest) to 100 (highest)
Processing Speed TMT-A | 11 months
  T-score, Trail Making Test: Part A (TMT; Reitan, 1971) Range: 0 (lowest) to 100 (highest)
Processing Speed Coding | 1 week
  T-score, Symbol Coding de la Brief Assessment of Cognition in Schizophrenia (BACS)(Keefe, 2004) Range: 0 (lowest) to 100 (highest)
Processing Speed Coding | 5 months
  T-score, Symbol Coding de la Brief Assessment of Cognition in Schizophrenia (BACS)(Keefe, 2004) Range: 0 (lowest) to 100 (highest)
Processing Speed Coding | 11 months
  T-score, Symbol Coding de la Brief Assessment of Cognition in Schizophrenia (BACS)(Keefe, 2004) Range: 0 (lowest) to 100 (highest)
Processing Speed FAS Word Fluency | 1 week
  T-score, FAS Word Fluency (Guilford, 1967) Range: 0 (lowest) to 100 (highest)
Processing Speed FAS Word Fluency | 5 months
  T-score, FAS Word Fluency (Guilford, 1967) Range: 0 (lowest) to 100 (highest)
Processing Speed FAS Word Fluency | 11 months
  T-score, FAS Word Fluency (Guilford, 1967) Range: 0 (lowest) to 100 (highest)
Processing Speed Semantic Word Fluency | 1 week
  T-score, Semantic Word Fluency (Guilford, 1967) Range: 0 (lowest) to 100 (highest)
Processing Speed Semantic Word Fluency | 5 months
  T-score, Semantic Word Fluency (Guilford, 1967) Range: 0 (lowest) to 100 (highest)
Processing Speed Semantic Word Fluency | 11 months
  T-score, Semantic Word Fluency (Guilford, 1967) Range: 0 (lowest) to 100 (highest)

SECONDARY OUTCOMES:
Psychopathology | 1 week
  qualitative nominal, Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS-PL-5)
Positive symptoms | 1 week
  qualitative ordinary Positive symptoms, Positive and Negative Syndrome Scale (PANSS) 7 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
Positive symptoms | 5 months
  qualitative ordinary Positive symptoms, Positive and Negative Syndrome Scale (PANSS)7 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
Positive symptoms | 11 months
  qualitative ordinary Positive symptoms, Positive and Negative Syndrome Scale (PANSS)7 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
Negative symptoms | 1 week
  qualitative ordinary Negative symptoms, of the "Positive and Negative Syndrome Scale (PANSS)".7 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
Negative symptoms | 5 months
  qualitative ordinary Negative symptoms, of the "Positive and Negative Syndrome Scale (PANSS)".7 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
Negative symptoms | 11 months
  qualitative ordinary Negative symptoms, of the "Positive and Negative Syndrome Scale (PANSS)".7 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
General psychopathology | 1 week
  qualitative ordinary Disorganization symptoms, Positive and Negative Syndrome Scale (PANSS)7 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
General psychopathology | 5 months
  qualitative ordinary Disorganization symptoms, Positive and Negative Syndrome Scale (PANSS) 16 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
General psychopathology | 11 months
  qualitative ordinary Disorganization symptoms, Positive and Negative Syndrome Scale (PANSS) 16 items, 1-7 scale (1:symptom is not present / 7:extrem presence of symptom); the number of symptoms that have punctuation of =4 or >4
IQ (WISC-V) | 1 week
  intelligence quotient, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014)
IQ | 1 week
  intelligence quotient, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012)(PANSS)
Family Psychiatric History | 1 week
  qualitative nominal, interview ad-hoc
socioeconomic status | 1 week
  qualitative nominal , interview ad-hoc
toxics | 1 week
  qualitative nominal , interview ad-hoc
toxics | 5 months
  qualitative nominal , interview ad-hoc
toxics | 11 months
  qualitative nominal , interview ad-hoc
Date of birth | 1 week
  qualitative nominal, ad-hoc
Sex | 1 week
  qualitative binary, ad-hoc
Obstetric Risk | 1 week
  Hollingshead and Redich Scale (1958)
Personal Psychiatric History | 1 week
  qualitative nominal , interview ad-hoc
Development History | 1 week
  qualitative nominal , interview ad-hoc
Medical History | 1 week
  qualitative nominal , interview ad-hoc
Psychiatric treatment | 1 week
  qualitative nominal , interview ad-hoc
Hospitalization | 1 week
  qualitative nominal , interview ad-hoc

OTHER OUTCOMES:
vocabulary (WISC-V) | 1 week
  T-score, vocabulary, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
vocabulary | 1 week
  T-score, vocabulary, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
similarities (WISC-V) | 1 week
  T-score, similarities, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
similarities | 1 week
  T-score, similarities, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
block design (WISC-V) | 1 week
  T-score, block design, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
block design | 1 week
  T-score, block design, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
matrix reasoning (WISC-V) | 1 week
  T-score, matrix reasoning, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
matrix reasoning | 1 week
  T-score, matrix reasoning, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
Figure Weights (WISC-V) | 1 week
  T-score, Figure Weights, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
Figure Weights | 1 week
  T-score, Figure Weights, /Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
verbal comprehension (WISC-V) | 1 week
  Index verbal comprehension Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 200 (highest)
verbal comprehension | 1 week
  Index verbal comprehension, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 200 (highest)
fluid reasoning (WISC-V) | 1 week
  Index fluid reasoning, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 200 (highest)
fluid reasoning | 1 week
  Index fluid reasoning, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 200 (highest)
Attention, omissions | 1 week
  T-scores, omissions, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, omissions | 5 months
  T-scores, omissions, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, omissions | 11 months
  T-scores, omissions, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, commissions | 1 week
  T-scores, commissions, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, commissions | 5 months
  T-scores, commissions, Continuous Performance Test - II (CPT-II; Rosvold, 1956)Range: 0 (lowest) to 100 (highest)
Attention, commissions | 11 months
  T-scores, commissions, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, reaction time | 1 week
  T-scores, hit reaction time, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, reaction time | 5 months
  T-scores, hit reaction time, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, reaction time | 11 months
  T-scores, hit reaction time, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, detectability | 1 week
  T-scores, detectability, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, detectability | 5 months
  T-scores, detectability, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, detectability | 11 months
  T-scores, detectability, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, variability | 1 week
  T-scores, variability, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, variability | 5 months
  T-scores, variability, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Attention, variability | 11 months
  T-scores, variability, Continuous Performance Test - II (CPT-II; Rosvold, 1956) Range: 0 (lowest) to 100 (highest)
Copy Visual Memory | 1 week
  T-score, copy, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991) Range: 0 (lowest) to 100 (highest)
Copy Visual Memory | 5 months
  T-score, copy, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991) Range: 0 (lowest) to 100 (highest)
Copy Visual Memory | 11 months
  T-score, copy, Rey-Osterrieth complex figure (HVLT-R; Brandt 1991) Range: 0 (lowest) to 100 (highest)
working memory direct digit (WISC-V) | 1 week
  T-score, direct Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
working memory direct digit | 1 week
  T-score, direct Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
working memory direct digit (WISC-V) | 5 months
  T-score, direct Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
working memory direct digit | 5 months
  T-score, direct Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
working memory direct digit (WISC-V) | 11 months
  T-score, direct Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
working memory direct digit | 11 months
  T-score, direct Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
working memory indirect digit (WISC-V) | 1 week
  T-score, indirect Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
working memory indirect digit | 1 week
  T-score, indirect Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
working memory indirect digit (WISC-V) | 5 months
  T-score, indirect Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) (Wechsler, 2014) Range: 0 (lowest) to 100 (highest)
working memory indirect digit | 5 months
  T-score, indirect Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
working memory indirect digit (WISC-V) | 11 months
  T-score, indirect Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) Range: 0 (lowest) to 100 (highest)(Wechsler, 2014)
working memory indirect digit | 11 months
  T-score, indirect Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
working memory growing digit (WISC-V) | 1 week
  T-score, growing Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) Range: 0 (lowest) to 100 (highest)(Wechsler, 2014)
working memory growing digit | 1 week
  T-score, growing Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
working memory growing digit (WISC-V) | 5 months
  T-score, growing Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) Range: 0 (lowest) to 100 (highest)(Wechsler, 2014)
working memory growing digit | 5 months
  T-score, growing Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
working memory growing digit (WISC-V) | 11 months
  T-score, growing Digits Test, Wechsler Intelligence Scale for Children-Five Edition (WISC-V) Range: 0 (lowest) to 100 (highest)(Wechsler, 2014)
working memory growing digit | 11 months
  T-score, growing Digits Test, Wechsler Intelligence Scale for Adults (WAIS-IV) (Wechsler, 2012) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT errors totals | 1 week
  T-score, errors totals Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT errors totals | 5 months
  T-score, errors totals Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT errors totals | 11 months
  T-score, errors totals Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage error | 1 week
  T-score, percentage error Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage error | 5 months
  T-score, percentage error Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage error | 11 months
  T-score, percentage error Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT perseverating responses | 1 week
  T-score, perseverating responses Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT perseverating responses | 5 months
  T-score, perseverating responses Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT perseverating responses | 11 months
  T-score, perseverating responses Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage perseverating errors | 1 week
  T-score, percentage perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage perseverating errors | 5 months
  T-score, percentage perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage perseverating errors | 11 months
  T-score, percentage perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT perseverating errors | 1 week
  T-score, perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT perseverating errors | 5 months
  T-score, perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT perseverating errors | 11 months
  T-score, perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT no perseverating errors | 1 week
  T-score, no perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT no perseverating errors | 5 months
  T-score, no perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT no perseverating errors | 11 months
  T-score, no perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage no perseverating errors | 1 week
  T-score, percentage no perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage no perseverating errors | 5 months
  T-score, percentage no perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)
executive functions, WSCT percentage no perseverating errors | 11 months
  T-score, percentage no perseverating errors Wisconsin Card Sorting Test (WCST; Heaton et al.,1981) Range: 0 (lowest) to 100 (highest)

CONTACTS AND LOCATIONS:
Overall Officials: Ester Camprodon Rosanas, Psychology, Principal Investigator — Hospital Sant Joan de Deu Barcelona
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT05405946/ICF_000.pdf